CLINICAL TRIAL: NCT03504072
Title: Risk of Tuberculosis and Infections in Spondyloarthritis Patients Treated With Tofacitinib in Bangladesh
Brief Title: Risk of Tuberculous and Other Infections in Patients of Spondyloarthritis Treated With Tofacitinib in Bangladesh
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Md. Nazrul Islam, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/547
Record Dates: First submitted 2018-03-29; First posted 2018-04-20 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Spondyloarthritis
Keywords: Etanercept; Infection; Tofacitinib; Tuberculosis; Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis; Infections; Tuberculosis | interventions — tofacitinib; Etanercept

STUDY DESIGN:
Intervention Model Description: Follow up period will be 9 months (visits 0, 1, 3, 6 and 9). Study subjects (87) will receive toficitinib (5 mg 12 hourly). Control patients will get eternacept (50 mg subcutaneously every 7 days interval for 1st month then 50 mg in 15 days interval for 2nd month then 50 mg every 21 days interval till final visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofacitinib 5mg (Active Comparator): tofacitinib 5 mg 12 hourly daily for 9 months. Evaluation schedule will be baseline, 1st month, 3rd months and 3 monthly for 9 months. relevant investigations will be done at each visit. occurrence of tuberculosis and infections will be recorded at follow up visits.
  Interventions: Drug: Tofacitinib 5 mg,
- Etanercept 50 mg (Active Comparator): Etanercept 50 mg subcutaneously every 7 days interval for 1st month then, Etanercept 50 mg in 15 days interval for 2nd month then 50 mg every 21 days interval for 9 months. Occurrence of tuberculosis and infections will be recorded at follow up visits.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Tofacitinib 5 mg, — tofacitinib 5 mg 12 hourly daily for 9 months
  Other Names: tofacitinib
  Arms: Tofacitinib 5mg
Drug: Etanercept — Etanercept 50 mg sc every 7 days interval in 1st month, every 15 days interval in 2nd month and then every 21 days interval from 3rd month onward upto 9 months
  Other Names: Etanercept 50 mg
  Arms: Etanercept 50 mg

SUMMARY:
Treatment failure of Spondyloarthropathies (SpA) leads to marked functional disability, higher rates of morbidity, mortality and poor quality of life. In TB endemic countries effective and safe drugs are to be in hand to manage this group of patients. The aim of this study will be to evaluation the risk of tuberculosis and other infections in refractory SpA patients treated with tofacitinib. After having consent 174 adults will be enrolled. Follow up period will be 9 months (visits 0, 1, 3, 6 and 9). Study subjects (87) will receive tofacitinib (5 mg 12 hourly). Control patients will get etanercept (50 mg subcutaneously every 7 days interval for 1st month then 50 mg in 15 days interval for 2nd month then 50 mg every 21 days interval till final visit.

Treatment efficacy assessment tool will be BASDAI, ASDAS-ESR, ASDAS-CRP and ASQoL for quality of life. Occurrences of tuberculosis and serious infection will be the primary end point of this study. The quantitative variables like ESR, CRP, BASDAI, ASDAS-ESR, ASDAS-CRP and ASQoL scores will be computed as mean and SD. Occurrences of TB and infection will be expressed in number and percentage. In between groups according to data distribution, students't test or ManWhitny U test will be done. The P value <0.05 will be considered significant. Each patient will enjoy every right to participate or refuse or even withdraw from the study at any point of time. Anonymity and data confidentiality will be maintained strictly. Ethical clearance will be obtained from Institutional Review Board (IRB) of BSMMU.

The expected utility of this study will be; a) reporting on occurrence of TB and other infections in SpA patients with tofacitinib and etanercept, b) if identified safe and effective physician can use the agents without fear, c) for dose spacing of etanercept the cumulative dose will be low might make the drug affordable and also reduce the risk of TB and other infections, d) for spaced follow up schedule there will be minimized physician visit, lab testing etc.

DETAILED DESCRIPTION:
Spondyloarthropathies (SpA) are non curable, diseases of young subjects, treatment failure leads to marked functional disability, higher rates of morbidity, mortality and poor quality of life. Effective drugs may not be safe in different geographic backgrounds. Bangladesh is a TB endemic country so patients are at risk of TB and other infections at background. The aim of this study will be to evaluation the risk of tuberculosis and other infections in refractory SpA patients treated with tofacitinib.

In this randomized clinical trial a total 174 adults will be enrolled from BSMMU and other hospitals of Dhaka city. The study period will be from January 2018 to December 2019. Subjects of both gender (≥18 years), who fulfil inclusion criteria will be enrolled after having informed written consent. Follow up period will be 9 months (visits 0, 1, 3, 6 and 9). Study subjects (87) will receive tofacitinib (5 mg 12 hourly). Control patients will get etanercept (50 mg subcutaneously every 7 days interval for 1st month then 50 mg in 15 days interval for 2nd month then 50 mg every 21 days interval till final visit. Demographics, clinical and lab information will be recorded in semi-structured schedule. Treatment efficacy assessment tool will be BASDAI, ASDAS-ESR, ASDAS-CRP and ASQoL for quality of life. Relevant lab test will be done at follow up visits. Side effects will be recorded in the research schedule. Occurrences of tuberculosis and serious infection will be the primary end point of this study. The demographics and categorical outcomes will be expressed in number and percentage. The quantitative variables like ESR, CRP, BASDAI, ASDAS-ESR, ASDAS-CRP and ASQoL scores will be computed as mean and SD. Occurrences of TB and infection will be expressed in number and percentage. Within group the quantitative data of baseline and of final visit will be analyzed using independent sample t test. In between groups according to data distribution, students't test or ManWhitny U test will be done. The P value <0.05 will be considered significant. Each patient will enjoy every right to participate or refuse or even withdraw from the study at any point of time. The study drugs are widely used agents in abroad for different rheumatic conditions having acceptable safety profile with efficacy as such there will be no extra risk of study subjects. Anonymity and data confidentiality will be maintained strictly. Ethical clearance will be obtained from Institutional Review Board (IRB) of BSMMU.

The expected utility of this study will be; a) reporting on occurrence of TB and other infections in SpA patients with tofacitinib and etanercept, b) if identified safe and effective physician can use the agents without fear, c) for dose spacing of etanercept the cumulative dose will be low might make the drug affordable and also reduce the risk of TB and other infections, d) for spaced follow up schedule there will be minimized physician visit, lab testing etc.

ELIGIBILITY:
Inclusion Criteria:

1. IBP criteria (4 out of 5 parameters present more than 3 months) Inflammatory back pain 1) Age of onset <45 yr 2) Insidious onset 3) Improvement with exercise 4) No improvement with rest 5) Pain at night (with improvement upon arising)
2. Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of > 4 (range, 0-10)
3. Failing to response to 2 NSAIDs in full therapeutic dose or withdrawal for intolerance in four consecutive weeks
4. Age > 18 years
5. Agreed to participate in the study

Exclusion Criteria:

1. Known case of allergic patients
2. Pregnancy
3. Patient with any active or history of any chronic or recurrent or serious or opportunistic infection/sepsis
4. Known case of chronic kidney disease (Cl cr <40 mL/minute)
5. Moderate to severe liver disease of any type
6. Lymphopenia (Lymphocyte <500 cells/mm3 of blood)
7. Neutropenia (Neutrophil <1000 cells/mm3 of blood)
8. Anaemia (Hb < 9 g/dl)
9. Who have been exposed to tuberculosis
10. Chest X-ray suggestive of pulmonary tuberculosis
11. Patients who do not want to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Tuberculosis | 9th months
  While on trial drug occurrence of tuberculosis either pulmonary or extra pulmonary

SECONDARY OUTCOMES:
improvement of disease activity measures of spondyloarthritis by >40% | at 9th month
  >40% improvement in at least 4 of the following 5 parameters: Patient global assessment, Pain, Function, Morning stiffness, Spinal mobility, C- reactive protein
  1. Patient global assessment
  2. Pain
  3. Function
  4. Morning stiffness
  5. Spinal mobility C- reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Shaikh A Al Mamun, MBBS, Study Chair — Member secretary
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No